CLINICAL TRIAL: NCT02277223
Title: Curcumin for Induction and Maintenance Therapy in Pediatric Ulcerative Colitis
Brief Title: Curcumin in Pediatric Ulcerative Colitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty to enroll patients
Sponsor: Schneider Children's Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Amit Assa, Pediatric Gastroenterologist, Schneider Children's Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PUCC 1
Record Dates: First submitted 2014-10-25; First posted 2014-10-28 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): In addition to induction therapy, patients will receive oral capsules of curcumin (Bara Herbs Inc): Weight<20kg: 1 gram, twice daily, 20-30 kg: 1.5 grams twice daily, weight>30kg: 2 grams twice daily. For Maintenance, in addition to oral 5-ASA maintenance treatment, responding patients will receive oral capsules of curcumin (Bara Herbs Inc): Weight<30kg: 500 milligram, twice daily, weight>30kg: 1 gram twice daily
  Interventions: Dietary Supplement: Curcumin
- Control (Placebo Comparator): In addition to induction and maintenance therapy, patients will receive matched oral placebo capsules for induction and maintenance (Bara Herbs Inc), twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin — Eligible patients will be randomized to either intervention of placebo groups. Randomization will be performed separately for patients receiving corticosteroids for induction in-order to ensure similar heterogeneity within groups. Induction: oral prednisone 1mg/kg up to 40 mg once daily for 2 weeks and then tapered down by 5 mg per week or 5-ASA 75 mg/kg/day divided to two doses. Maintenance: 5-ASA 75 mg/kg/day divided to two doses.
  Patients receiving corticosteroids for induction, whose PUCAI is >35 points at 2 weeks will be regarded as treatment failure. Patients receiving 5-ASA for induction with "induction treatment failure" will be re-randomized to receive oral corticosteroids induction with or without curcumin.
  Other Names: Tumeric
  Arms: Interventional
Drug: Placebo — Eligible patients will be randomized to either intervention of placebo groups. Randomization will be performed separately for patients receiving corticosteroids for induction in-order to ensure similar heterogeneity within groups. Induction: oral prednisone 1mg/kg up to 40 mg once daily for 2 weeks and then tapered down by 5 mg per week or 5-ASA 75 mg/kg/day divided to two doses. Maintenance: 5-ASA 75 mg/kg/day divided to two doses.
  Patients receiving corticosteroids for induction, whose PUCAI is >35 points at 2 weeks will be regarded as treatment failure. Patients receiving 5-ASA for induction with "induction treatment failure" will be re-randomized to receive oral corticosteroids induction with or without curcumin.
  Other Names: Matched placebo
  Arms: Control

SUMMARY:
Background: Curcumin in an active phytochemical substance, used as part of the human diet, that has anti-inflammatory and anti-oxidative properties which were demonstrated in multiple experimental models of colitis including a positive effect on maintenance of remission in adult ulcerative colitis (UC) patients. Objectives: To examine the effect of curcumin as complementary medication in induction and maintenance therapy in pediatric patients with mild to moderate ulcerative colitis. Design: A prospective, randomized, placebo-controlled study. Setting: Pediatric gastroenterology centers. Participants: Children 6 year to 18 years who are diagnosed with mild to moderate UC and are planned to receive either 5-ASA or corticosteroids induction treatment. Main outcome measures: Disease activity defined by the Pediatric Ulcerative Colitis Activity Index (PUCAI) at 2 weeks and 6 months. Secondary outcome measures: Effect of curcumin treatment on serum inflammatory markers, calprotectin and fecal microbiota. Data analysis: Data will be collected and analyzed using SPSS (version 21.0, SPSS, Inc., Chicago, IL, USA). Fisher's exact test will be used to explore univariate associations between primary outcomes and categorical variables. Associations of continues variables with primary outcome measures will be examined using ANOVA with repeated measures. P-values <0.05 will be considered significant.

DETAILED DESCRIPTION:
Clinical efficacy of induction and maintenance medications in pediatric UC is limited with a cumulative long-term risk of 20%-30% for colectomy. Remission rates following induction with corticosteroids and 5-amino-salicylic acid (5-ASA) range from 20% to 50%. 5-ASA is still regarded as first line induction and maintenance therapy for mild to moderate UC in both children and adults. 5-ASA is also indicated for maintenance therapy following successful induction with corticosteroids for moderate to severe disease. Still, steroid free clinical remission at 1 year under 5-ASA maintenance therapy is reported to range from 40% to 50%. Management of recurrent flares while taking 5-ASA medications involves repeated courses of corticosteroids and changing therapeutic regimes to include more potent medications such as thiopurines which carry an increased risk for significant adverse effects. Hence, improving efficacy of induction and maintenance treatment is of critical importance. Curcumin, an active phytochemical substance with anti-inflammatory properties was studied extensively in-vitro and in experimental models of colitis. In the only randomized controlled trial, performed in adults with quiescent disease, curcumin was shown to be an effective concomitant treatment (along with 5-ASA) for maintenance of remission. Therefore, our aim is to assess the efficacy of concomitant curcumin maintenance therapy for induction and maintenance therapy in pediatric UC patients with mild to moderate in a prospective randomized, placebo controlled trial. We hope that this study will further contribute to the understanding of the potential benefits of curcumin in pediatric UC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of UC, established by the presence of accepted clinical, radiologic, endoscopic and histologic criteria.
2. Age: 6 - 18 years (inclusive).
3. PUCAI 10-65 at enrollment
4. Negative stool culture, parasites and clostridium toxin
5. Ability and acceptance to participate in the study and follow study procedures, as evidenced by a parent/legal guardian signing a written informed consent and the child providing assent.

Exclusion Criteria:

1. Acute severe UC (PUCAI>65 points) requiring IV corticosteroids.
2. History of two relapses or more on 5-ASA treatment.
3. Pregnancy
4. Sepsis or active bacterial infection
5. Fever >38.5 degrees.
6. Patients whose disease is confined to the rectum (i.e. proctitis).
7. Patients with crohn's colitis or with IBD type unclassified (IBD-U) according to Montreal classification.
8. Rectal therapies (suppositories, foams, enemas etc) of all kind are allowed if the dose and frequency has remained stable during the previous 14 days prior to the screening visit.
9. Known allergy to 5ASA, salicylates, or aminosalicylates.
10. History of recurrent pancreatitis.
11. Existence of current renal disease, or a screening blood urea nitrogen (BUN) or creatinine value that is > 1.5 times the upper limit of the age appropriate normal.

    -

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
A change in disease activity, defined by PUCAI at 2 weeks and 6 months | 6 months

SECONDARY OUTCOMES:
Sustained clinical remission, 2 weeks and 6 months | 6 months
Medication associated adverse events | 6 months
Time to relapse | 6 months
The need for further medical interventions (e.g topical 5-ASA) during the maintenance phase | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amit Assa, MD, Principal Investigator — Schneider Children's Medical Center
Locations (1):
- Schneider Medical Center, Petah Tikva, Israel